CLINICAL TRIAL: NCT04320771
Title: Investigation of Pharmacokinetics, Safety and Tolerability of Neladenoson Bialanate in Male and Female Subjects With Renal Impairment and in Age-, Gender-, and Weight-matched Healthy Subjects Following a Single Oral Dose of 10 mg Neladenoson Bialanate Given as IR Tablet in a Single-center, Nonrandomized, Non-controlled, Non-blinded, Study With Group Stratification
Brief Title: Study on the Safety of Neladenoson Bialanate, How it is Tolerated and the Way the Body Absorbs, Distributes and Gets Rid of the Study Dug Given as a Single Oral Dose of 10 mg Immediate Release Tablet in Participants With Renal Impairment and Healthy Participants Matched for Age-, Gender-, and Weight
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Termination of the development project for Neladenoson bialanate
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15138; 2017-000795-28 (EudraCT Number)
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Pharmacology, Clinical
MeSH Terms: interventions — neladenoson bialanate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neladenoson bialanate, mild renal impairment (Experimental): Subjects with eGFR ≥60 - <90 mL/min/1.73 received a single immediate-release (IR) tablet dose of 10 mg of neladenoson bialanate in the fasted state
  Interventions: Drug: Neladenoson bialanate (BAY 1067197)
- Neladenoson bialanate, moderate renal impairment (Experimental): Subjects with eGFR ≥30 - <60 mL/min/1.73 received a single IR tablet dose of 10 mg of neladenoson bialanate in the fasted state
  Interventions: Drug: Neladenoson bialanate (BAY 1067197)
- Neladenoson bialanate, severe renal impairment (Experimental): Subjects with eGFR <30 mL/min/1.73 received a single IR tablet dose of 10 mg of neladenoson bialanate in the fasted state
  Interventions: Drug: Neladenoson bialanate (BAY 1067197)
- Neladenoson bialanate, control group (Experimental): Healthy subjects matched for age, gender and body weight received a single IR tablet dose of 10 mg neladenoson bialanate in the fasted state
  Interventions: Drug: Neladenoson bialanate (BAY 1067197)

INTERVENTIONS:
Drug: Neladenoson bialanate (BAY 1067197) — 10 mg as a single IR tablet dose. Active metabolite: BAY 84-3174

SUMMARY:
Neladenoson bialanate is currently under clinical development for a condition in which the heart has trouble pumping blood through the body (chronic heart failure). Renal impairment which co-occurs in patients with heart failure is a common condition in which the kidneys are not filtering the blood as well as they should. The goal of the study is to learn more about the safety of neladenoson bialanate, how it is tolerated and the way the body absorbs, distributes and excretes the study dug given as a single oral dose of 10 mg immediate release tablet in participants with renal impairment and healthy participants matched for age-, gender-, and weight

DETAILED DESCRIPTION:
Study was originally designed with 4 arms (normal renal function, mild, moderate, and severe renal impairment), however as the study was prematurely terminated, there was no participant with normal renal function enrolled

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Male or female White subjects (women without childbearing potential), aged 18 to 79 years (inclusive), body mass index 18 to 34 kg/m² (both inclusive)

Subjects with renal impairment:

* Estimated glomerular filtration rate (eGFR) <90 mL/min/1.73 m² determined from serum creatinine 2-14 days prior to dosing using the Modification of Diet in Renal Disease equation
* Stable renal disease, i.e. a serum creatinine value determined at least 3 months before the pre-study visit should not vary by more than 25% from the serum creatinine value determined at the pre-study visit.

Healthy subjects:

* Age-, weight- and gender matched healthy subjects

Exclusion Criteria:

* An anatomical abnormality of the gut (e.g. gut surgery, continent ileostomy) that could affect the retention times of the drug in the stomach/gut adversely
* Gastric vagotomy or other condition that might adversely affect the gastric pH level
* Pancreatic dysfunction/insufficiency
* Febrile illness within 1 week prior to admission to study center
* Use of the following co-medications

From 2 weeks before administration until end of follow-up:

* Cytochrome P450 (CYP)3A4 inhibitors (Of note: grapefruit is a strong CYP3A4 inhibitor)
* CYP3A4 inducers
* CYP2C8 inhibitors (Of note: clopidogrel is a strong CYP2C8 inhibitor)
* Theophylline

On the day of dosing with neladenoson bialanate:

* Drugs that undergo significant systemic metabolism over gut wall uridine diphosphate-glucuronosyltransferase 1A1 (UGT1A1) substrates (e.g. irinotecan)
* Major breast cancer resistance protein (BCRP) substrates
* Regular daily consumption of more than 1 L - Plasmapheresis within 4 weeks before study drug administration
* Therapies (e.g. physiotherapy, acupuncture, etc.) within 1 week before study drug administration
* History of relevant and not cured cardiac rhythm disorders (i.e. Wolff-Parkinson-White syndrome, intermittent second- or third-degree AV block)
* Positive urine drug screening
* Subjects tested to be positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Cmax for BAY 84-3174 | Pre-dose up to approximately 6 weeks after dosing
  Maximum observed drug concentration in measured matrix after single dose administration
AUC for BAY 84-3174 | Pre-dose up to approximately 6 weeks after dosing
  Area under the concentration vs. time curve from zero to infinity after single dose administration
Cmax,norm for BAY 84-3174 | Pre-dose up to approximately 6 weeks after dosing
  Cmax divided by dose per body weight after single dose administration
AUCnorm for BAY 84-3174 | Pre-dose up to approximately 6 weeks after dosing
  AUC divided by dose per body weight after single dose administration
Cmax,u for BAY 84-3174 | Pre-dose up to approximately 6 weeks after dosing
  Cmax of unbound drug after single dose administration
AUCu for BAY 84-3174 | Pre-dose up to approximately 6 weeks after dosing
  AUC of unbound drug after single dose administration
fu for BAY 84-3174 | At 4 hours after dosing
  Fraction of free (unbound) drug in plasma or serum after single dose administration

SECONDARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAEs) | Up to approximately 6 weeks after dosing

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - APEX GmbH, München, Bavaria
  - CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/